CLINICAL TRIAL: NCT01285635
Title: A Phase II of AT-101 in Combination With Docetaxel in Patients With Recurrent, Locally Advanced or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: A Study of AT-101 in Combination With Docetaxel in Squamous Cell Carcinoma Of The Head and Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug is no longer manufactured
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2010.031; HUM00040432 (Other: University of Michigan IRB Number)
Record Dates: First submitted 2011-01-20; First posted 2011-01-28 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck (SCCHN)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — gossypol acetic acid; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Docetaxel Alone (Active Comparator)
  Interventions: Drug: Docetaxel
- Pulse Dose AT-101 Arm (Experimental)
  Interventions: Drug: AT-101; Drug: Docetaxel
- Metronomic AT-101 Arm (Experimental)
  Interventions: Drug: AT-101; Drug: Docetaxel

INTERVENTIONS:
Drug: AT-101 — Pulse Dose: AT-101 dose of 40 mg b.i.d. on days 1-3 Metronomic Dose: AT-101, 20 mg daily, days 1-14
  Arms: Metronomic AT-101 Arm; Pulse Dose AT-101 Arm
Drug: Docetaxel — Docetaxel 75 mg/m2 on Cycle Day 1

SUMMARY:
This study will examine the effects of an investigational drug called AT-101 in combination with an FDA approved cancer drug called Docetaxel. It is hoped that AT-101 will help the Docetaxel to have a better effect in slowing or stopping cancer cell growth. This study will help the researchers learn what effects, if any, the combination of AT-101 and Docetaxel has on your cancer. For instance, will the combination cause your tumor(s) to shrink or stop growing? The researchers will also learn about the safety of the combination of AT-101 and Docetaxel. For instance, are there any side effects? If so, what kind of side effects does the combination cause? How severe are the side effects, and how often do they occur?

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females at least 18 years old.
2. Histologically or cytologically confirmed diagnosis of SCCHN (Squamous Cell Carcinoma of the Head and Neck).
3. Stage IVC (metastatic), or advanced, locally recurrent SCCHN not amenable to surgery or palliative radiotherapy.
4. Presence of measurable disease as defined by RECIST (Response Evaluation Criteria in Solid Tumors)

   a. If the only site of measurable disease for this study is within a prior field of irradiation, then the sum of the longest diameter (SLD) of that lesion must have increased by at least 20% from the prior treatment nadir
5. Received no more than two prior systemic chemotherapeutic regimen for SCHNN in the locally advanced or metastatic setting and have relapsed after or be refractory to therapy

   * Systemic therapies given in the adjuvant setting or with chemoradiotherapy are counted only if the patient relapses after 6 months of the last cycle of chemotherapy or the completion of radiation
   * Included as systemic chemotherapy regimens (but not limited to) are patients who may have received erlotinib (Tarceva®) or another EGFR inhibitor. Previous treatment with paclitaxel (but not docetaxel) is permitted.
6. ECOG performance status ≤ 1 (Appendix 2)
7. Expected survival of at least 3 months
8. Adequate liver and renal and bone marrow function as indicated by:

   * Serum creatinine ≤ 2.0 times the upper limit of normal, AND
   * Serum albumin ≥ 3.0 gm/dL, AND
   * Total bilirubin ≤ 1.0 times the upper limit of normal, AND
   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN) for the testing laboratory. Note: For patients with alkaline phosphatase ≥ 2.5 x ULN, the AST and ALT must be ≤ 1.5 x ULN
   * Hemoglobin ≥ 9 g/dL (may be post-transfusion);
   * Platelet count ≥ 100 x103 cells/mm3
   * Neutrophil count ≥1500 cells/mm3
9. Negative pregnancy test for females of childbearing potential
10. Willingness to use contraception by a method that is deemed effective by the Investigator by both males and female patients of childbearing potential (postmenopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least 30 days following the last dose of AT-101
11. Ability to understand and the willingness to sign a written informed consent form; the consent form must be signed by the patient prior to any study-specific procedures
12. Willingness and ability to comply with study procedures and follow-up examination

Exclusion Criteria:

1. Pregnant or nursing women.
2. Prior docetaxel treatment for SCCHN in the metastatic setting.
3. Treatment of SCCHN with chemotherapy within 28 days of the first dose of study treatment. Acute toxicities from prior therapy must have resolved to Grade ≤ 1. Patients whose disease responded to the most recently administered prior regimen must have documented progression of disease subsequent to that regimen, to be eligible.
4. Treatment with monoclonal antibody (e.g., VEGF or EGFR targeting antibody) within 45 days prior to the first dose of study treatment. Acute toxicities from prior therapy must have resolved to Grade ≤ 1. Patients whose disease responded to the most recently administered prior regimen must have documented progression of disease subsequent to that regimen, to be eligible.
5. Treatment of SCCHN with radiotherapy within 14 days of the first dose of study treatment. Prior radiotherapy is permissible only if the lesions used for determination of disease activity (i.e., target lesions) were not previously irradiated, or have increased in size since the completion of radiotherapy, and the patient has fully recovered from any toxicity of the radiotherapy.
6. Treatment of SCCHN with erlotinib within 14 days of the first dose of study treatment. Acute toxicities from prior therapy must have resolved to Grade ≤ 1. Patients whose disease responded to the most recently administered prior regimen must have documented progression of disease subsequent to that regimen, to be eligible.
7. Any concurrent therapy intended to treat SCCHN.
8. Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
9. Symptomatic hypercalcemia or hypercalcemia that is > Grade 2.
10. Participation in any investigational drug study within 28 days prior to study treatment. (Patient must have recovered from all acute effects of previously administered investigational agents).
11. Active secondary malignancy or history of other malignancy within the last five years (patients who have been disease-free for five years, or have a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible).
12. Active symptomatic fungal, bacterial and/or viral infection including active HIV. Note: protocol does not require screening for viruses; however, patients with known active infections are excluded.
13. Patients who are contraindicated for treatment with docetaxel.
14. Have malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, ulcerative colitis, inflammatory bowel disease, partial or complete small bowel obstruction.
15. Uncontrolled CNS (Central Nervous System) metastases. Patients with known, previously treated CNS metastases are eligible if they are neurologically stable, as per the investigating physician's clinical assessment, and do not require steroids at the time of study entry.
16. Prior use of gossypol or AT-101, or known hypersensitivity to gossypol or AT-101.
17. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
18. Any patient being treated for acute deep vein thrombosis or patients with a history of recurrent deep vein thrombosis independent of treatment with anticoagulation.
19. Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Worden, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients will receive arm specific therapy for the first two cycles, then all patients will be switched into the metronomic AT-101 arm for up to 10 cycles.
Groups:
- Docetaxel Then Metronomic AT-101: Docetaxel (75 mg/m2 on Cycle Day 1) for 2 weeks then AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles.
- Pulse AT-101 Then Metronomic AT-101: AT-101 (40 mg b.i.d. on days 1-3) then AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles.
- Metronomic AT-101 Arm: AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles.
Period: First Intervention (2 Weeks)
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Started | 13 | 11 | 11
Completed | 13 | 11 | 11
Not Completed | 0 | 0 | 0
Period: Second Intervention (10, 3 Week Cycles)
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Started | 13 | 11 | 11
Completed | 13 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm | Total
Number analyzed (Participants) | 13 | 11 | 11 | 35
Age, Continuous [Mean (Full Range); unit: years] | 56 [35 to 75] | 56 [38 to 67] | 59 [41 to 74] | 56 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 11 | 9 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Complete Response (CR) and Partial Response (PR)
Description: The primary objective is to estimate the proportion of patients with a complete response (CR) and partial response(PR) defined by RECIST (Response Evaluation Criteria in Solid Tumors). CR is defined as the disappearance of all target lesions and PR is defined as at least a 20% decrease in the sum of the longest diameter of target lesions.
Time Frame: 12 months
Measure: Number; unit: Patients
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Number analyzed (Participants) | 13 | 11 | 11
Patients
  Number of Patients with a CR | 0 | 0 | 0
  Number of Patients with a PR | 1 | 1 | 2

2. Secondary Outcome: Median Duration of Response For All Groups Combined
Time Frame: 3 years
Population: All patients on study
Measure: Median (Full Range); unit: months
Groups:
- Docetaxel and AT-101: Patients all receive Docetaxel 75mg/m^2 on Day 1. Patients will receive AT-101 on one of the following arms:
  Arm A: Docetaxel alone for two weeks, then AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles.
  Arm B: AT-101 (40 mg b.i.d. on days 1-3) then AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles
  Arm C: AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles.
Arm/Group | Docetaxel and AT-101
Number analyzed (Participants) | 35
months | 1.9 [0.2 to 16]

3. Secondary Outcome: Incidence of Grade 3 and 4 Toxicities by Arm
Description: Measure the grade III/IV toxicities experienced by patients with advanced, locally recurrent, or metastatic SCCHN
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Number analyzed (Participants) | 13 | 11 | 11
participants
  Fatigue | 2 | 1 | 0
  Anorexia | 1 | 2 | 1
  Nausea | 1 | 5 | 0
  Bowel Obstruction | 1 | 0 | 1
  Hematologic | 14 | 8 | 4
  Infectious | 4 | 0 | 1
  Respiratory | 1 | 0 | 3
  Edema | 0 | 2 | 1
  Other | 1 | 2 | 1

4. Secondary Outcome: Median Overall Survival in Months
Time Frame: 3 Years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pulse AT-101 Then Metronomic AT-101; Metronomic AT-101 Arm: AT-101 (20mg daily days 1-14) and Docetaxel (75 mg/m2 on Cycle Day 1) for up to 10 cycles.
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Number analyzed (Participants) | 13 | 11 | 11
months | 8.3 [5.5 to 9.9] | 4.9 [2.1 to 24] | 4.9 [2.7 to 13.7]

5. Secondary Outcome: Median Progression Free Survival in Months
Description: Progression is defined, by RECIST (Response Evaluation Criteria in Solid Tumors), as at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: 3 Years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Number analyzed (Participants) | 13 | 11 | 11
months | 4.5 [2.6 to 9.9] | 2.8 [1.2 to 5.9] | 4.2 [1.2 to 5.6]

ADVERSE EVENTS:
Arm/Group | Docetaxel Then Metronomic AT-101 | Pulse AT-101 Then Metronomic AT-101 | Metronomic AT-101 Arm
Serious Adverse Events (participants affected / at risk) | 6/13 | 7/11 | 6/11
Other Adverse Events (participants affected / at risk) | 12/13 | 11/11 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Then Metronomic AT-101 (N=13) | Pulse AT-101 Then Metronomic AT-101 (N=11) | Metronomic AT-101 Arm (N=11)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Jejunal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Periorbital infection (Infections and infestations) | 1 | 0 | 0
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 2 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Death NOS (General disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 0 | 1
Hypotension (Cardiac disorders) | 0 | 0 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Then Metronomic AT-101 (N=13) | Pulse AT-101 Then Metronomic AT-101 (N=11) | Metronomic AT-101 Arm (N=11)
Agitation (Psychiatric disorders) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 3 | 1
Alkaline phosphatase increased (Investigations) | 3 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 8 | 9 | 7
Anorexia (Metabolism and nutrition disorders) | 4 | 6 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Blurred vision (Eye disorders) | 1 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 1
Cholesterol high (Investigations) | 2 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1
Creatinine increased (Investigations) | 3 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 4
Dizziness (Ear and labyrinth disorders) | 3 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
Edema limbs (General disorders) | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Eye disorders - Other (Eye disorders) | 2 | 0 | 1
Fatigue (General disorders) | 8 | 7 | 5
Fever (General disorders) | 1 | 2 | 1
Flushing (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Genital edema (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 5 | 5
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 4 | 3
Hypotension (Cardiac disorders) | 1 | 1 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
INR increased (Investigations) | 1 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Laryngeal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lymph node pain (Vascular disorders) | 1 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 5 | 5 | 5
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 6 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 2 | 1
Otitis externa (Ear and labyrinth disorders) | 1 | 0 | 0
Pain (General disorders) | 3 | 2 | 2
Pain in extremity (General disorders) | 2 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 2 | 2 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash pustular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Scleral disorder (Eye disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Sore throat (Gastrointestinal disorders) | 1 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 1 | 0 | 0
Tremor (General disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Vascular disorders - Other (Vascular disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 0
Watering eyes (Eye disorders) | 1 | 0 | 0
Weight loss (General disorders) | 3 | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
White blood cell decreased (Blood and lymphatic system disorders) | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Chills (General disorders) | 0 | 2 | 0
Edema face (General disorders) | 0 | 1 | 1
Facial pain (General disorders) | 0 | 1 | 2
Gingival pain (General disorders) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypertension (Cardiac disorders) | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injection site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Malaise (General disorders) | 0 | 1 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0
Sinus pain (General disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Cognitive disturbance (Psychiatric disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Eyelid function disorder (Eye disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Flu like symptoms (Infections and infestations) | 0 | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Hot flashes (Endocrine disorders) | 0 | 0 | 1
Hyperhidrosis (Endocrine disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lethargy (General disorders) | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Otitis media (Ear and labyrinth disorders) | 0 | 0 | 1
Salivary gland infection (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Surgical and medical procedures - Other (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes